CLINICAL TRIAL: NCT00933647
Title: Effects of Yerba Mate and Green Tea Consumption on Cardiovascular Risk Factors in Dyslipidemic and Overweight Subjects
Brief Title: Cardioprotective Effects of Green Tea Versus Maté Intake
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Bruna Pontin, Instituto de Cardiologia / Fundação Universitária de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Projeto Chimarrão
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Dyslipidemia; Inflammation; Obesity
Keywords: Camellia sinensis; Ilex paraguariensis; Green tea; Yerba mate tea; Maté; Dyslipidemia; Inflammation; Obesity
MeSH Terms: conditions — Dyslipidemias; Inflammation; Obesity | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yerba Mate Tea (Experimental): Subjects will drink 1000ml/day of yerba mate tea for 8 weeks.
  Interventions: Dietary Supplement: Yerba Mate Tea
- Green Tea (Active Comparator): Subjects will drink 1000ml/day of green tea for 8 weeks.
  Interventions: Dietary Supplement: Green tea
- Apple Tea (Placebo Comparator): Subjects will drink 1000ml/day of apple tea for 8 weeks.
  Interventions: Dietary Supplement: Apple tea

INTERVENTIONS:
Dietary Supplement: Yerba Mate Tea — Before and after 8 weeks, serum lipids, C-reactive protein and fibrinogen will be measured. They will also be tested for glycemia, insulin, aminotransferases, bilirubin. Anthropometric measurements will be also performed at week 0 and 8. The subjects will receive instructions to maintain their usual dietary intake and normal physical activity.
  Arms: Yerba Mate Tea
Dietary Supplement: Green tea — Before and after 8 weeks, serum lipids, C-reactive protein and fibrinogen will be measured. They will also be tested for glycemia, insulin, aminotransferases, bilirubin. Anthropometric measurements will be also performed at week 0 and 8. The subjects will receive instructions to maintain their usual dietary intake and normal physical activity.
  Arms: Green Tea
Dietary Supplement: Apple tea — Before and after 8 weeks, serum lipids, C-reactive protein and fibrinogen will be measured. They will also be tested for glycemia, insulin, aminotransferases, bilirubin. Anthropometric measurements will be also performed at week 0 and 8. The subjects will receive instructions to maintain their usual dietary intake and normal physical activity.
  Arms: Apple Tea

SUMMARY:
The investigators aim to study the effects of green tea and maté consumption on lipid and inflammatory profiles in dyslipidemic and overweight subjects.

DETAILED DESCRIPTION:
Recommendations of lifestyle and dietary content changes are often made for primary prevention and improvement of many health conditions, including cardiovascular disease. For centuries, green tea (Camellia sinensis) has been linked to good health. Nowadays, it is considered a functional food because of its physiological benefits, mainly in terms of cardiovascular prevention. Green tea is considered one of the best sources of phenolic compounds, which possess antioxidant properties that may contribute to a reduction in the risk of cardiovascular disease. Lesser-known worldwide, but widely consumed in southern Latin America countries, yerba mate tea (Ilex paraguariensis) is also a good source of phenolic compounds. The antioxidant capacity of green tea has been extensively studied; however, few studies have reported that the antioxidant properties of maté tea is even greater than green tea. For this reason, the present study aims to compare the possible effects of the oral ingestion of maté and green tea on the lipid and inflammatory profiles in a southern Brazilian population.

ELIGIBILITY:
Inclusion Criteria:

* age 35-60 years
* non-treated dyslipidemia (TC > 200mg/dL and/or TG > 150 mg/dL and/or HDL-c < 40 mg/dL for men and 50mg /dL for women)
* BMI 25-35 Kg/m²

Exclusion Criteria:

* use or indication for use of lipid-lowering agents and/or vitamin supplement
* non-steroids anti inflammatory use
* hormone replacement therapy
* contraceptive use
* pregnancy
* nursing
* unexplained weight loss (>2 Kg) 2 months before the study
* altered hepatic function
* those who do not sign the informed consent

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of lipid (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total cholesterol / HDL-cholesterol ratio) and inflammatory profiles (C- reactive protein and fibrinogen). | 8 weeks

SECONDARY OUTCOMES:
Decreases in body weight, body mass index, body fat ratio, abdominal and waist circumferences and waist to hip ratio. Changes in glucose and insulin will also be evaluated. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vera Lúcia Portal, PhD, Study Director — Instituto de Cardiologia / Fundação Universitária de Cardiologia; Bruna Pontin, MD, Principal Investigator — Instituto de Cardiologia / Fundação Universitária de Cardiologia; Lúcia Campos Pellanda, PhD, Study Director — Instituto de Cardiologia / Fundação Universitária de Cardiologia
Locations (1):
- Instituto de Cardiologia / Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Balsan G, Pellanda LC, Sausen G, Galarraga T, Zaffari D, Pontin B, Portal VL. Effect of yerba mate and green tea on paraoxonase and leptin levels in patients affected by overweight or obesity and dyslipidemia: a randomized clinical trial. Nutr J. 2019 Jan 19;18(1):5. doi: 10.1186/s12937-018-0426-y. PMID 30660196